

Department of Social Sciences & Health Policy

# PREPARE TO CARE, A SUPPORTED SELF-MANAGEMENT INTERVENTION FOR HEAD AND NECK CANCER CAREGIVERS

Informed Consent Form to Participate in Research Chandylen Nightingale, PhD, MPH, Principal Investigator

# Introduction

You are invited to be in a research study. Research studies are designed to gain scientific knowledge that may help other people in the future. You are being asked to take part in this study because you are receiving radiation treatment for head and neck cancer and have a loved one providing care for you. Your participation is voluntary. Please take your time in making your decision as to whether or not you wish to participate. Ask your study doctor or the study staff to explain any words or information contained in this informed consent document that you do not understand. You may also discuss the study with your friends and family.

## WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to determine our ability to recruit caregivers of patients with head and neck cancer being treated with radiotherapy to a study that includes a kit, *Prepare to Care*, which may increase knowledge about head and neck cancer and enhance stressmanagement skills. We will also determine how many caregivers continued to use the kit during the study period, what caregivers liked and disliked about the kit, and make modifications to improve the *Prepare to Care* kit. In this study we also want to look at our ability to recruit a waitlist control group of caregivers, that is, caregivers of patients with head and neck cancer being treated with radiotherapy that receive the *Prepare to Care* Kit after the study has ended. Control groups are used in research to see if the intervention being studied really does have an effect.

## HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

40 caregivers and 40 patients from this research site will take part in this study.

#### WHAT IS INVOLVED IN THE STUDY?

If you take part in this study, we will collect basic information including demographics and clinical information (related to your diagnosis and treatment for head and neck cancer) from your medical record.

# HOW LONG WILL I BE IN THE STUDY?

You will be in the study for approximately 12-13 weeks, depending on the duration of your RT treatment. This includes the duration of your radiation treatment, typically lasting up to 6-7 weeks, and one follow up study visit which will take place 6 weeks after you have completed radiation treatment.

You can stop participating at any time. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or


Adult Consent Form



safety consequences. There are no consequences to withdrawing from this study.

# WHAT ARE THE RISKS OF THE STUDY?

The risk of harm or discomfort that may happen as a result of taking part in this research study is not expected to be more than in daily life or from routine physical or psychological examinations or tests. You should discuss the risk of being in this study with the study staff.

Taking part in this research study may involve providing information that you consider confidential or private. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe.

## ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

You are not expected to receive any direct benefit from taking part in this research study. We hope the information learned from this study will benefit other people in the future. There may or may not be direct benefit to your loved one.

#### WHAT OTHER CHOICES ARE THERE?

This is not a treatment study. Your alternative is to not participate in this study.

# WHAT ARE THE COSTS?

There are no costs to you for taking part in this study. Costs for your regular medical care, which are not related to this study, will be your own responsibility.

# WILL YOUR RESEARCH RECORDS BE CONFIDENTIAL?

The results of this research study may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed unless it is authorized by you, required by law, or necessary to protect the safety of yourself or others. There is always some risk that even de-identified information might be re-identified.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects.

The Certificate cannot be used to refuse a request for information from personnel of the United States federal or state government agency sponsoring the project that is needed for auditing or


Adult Consent Form



program evaluation by the National Cancer Institute which is funding this project or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it.

The Certificate of Confidentiality will not be used to prevent disclosure as required by federal, state, or local law of harm to self or others. The Certificate of Confidentiality will not be used to prevent disclosure for any purpose you have consented to in this informed consent document including all research data.

Participant information may be provided to Federal and other regulatory agencies as required. The Food and Drug Administration (FDA), for example, may inspect research records and learn your identity if this study falls within its jurisdiction.

# WILL YOU BE PAID FOR PARTICIPATING?

You will receive no payment or other compensation for taking part in this study.

## WHO IS SPONSORING THIS STUDY?

This study is being sponsored by the National Cancer Institute and the Comprehensive Cancer Center of Wake Forest Baptist Medical Center. The sponsor is providing money or other support to Wake Forest University Health Sciences to help conduct this study. The researchers do not, however, hold a direct financial interest in the sponsor or the intervention (*Prepare to* Care kit) being studied.

You do not give up any legal rights as a research participant by signing this consent form. For more information on medical treatment for research related injuries or to report a study related illness, adverse event, or injury you should call Dr. Chandylen Nightingale.

## WHAT ABOUT MY HEALTH INFORMATION?

In this research study, any new information we collect from you about your health or behaviors is considered <u>Protected Health Information</u>. The information we will collect for this research study includes: age, gender, information about your cancer diagnosis and treatment plan.

If this research study involves the diagnosis or treatment of a medical condition, then Protected Health Information collected from you during this study may be placed in your medical record, and may be used to help treat you, arrange payment for your care, or assist with Medical Center operations.

We will make every effort to keep your Protected Health Information private. We will store


Adult Consent Form



records of your Protected Health Information in a cabinet in a locked office or on a password protected computer.

Your personal health information and information that identifies you ("your health information") may be given to others during and after the study. This is for reasons such as to carry out the study, to determine the results of the study, to make sure the study is being done correctly, to provide required reports and to get approval for new products.

Some of the people, agencies and businesses that may receive and use your health information are members of the study team; the Institutional Review Board; and representatives of Wake Forest University Health Sciences and North Carolina Baptist Hospital.

If required by law or court order, we might also have to share your Protected Health Information with a judge, law enforcement officer, government agencies, or others. If your Protected Health Information is shared with any of these groups it may no longer be protected by federal or state privacy rules.

Any Protected Health Information collected from you in this study that is maintained in the research records will be kept for at least three years after the study is finished. You will not be able to obtain a copy of your Protected Health Information in the research records until all activities in the study are completely finished.

You can tell **Dr. Chandylen Nightingale, PhD, MPH** that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:

Chandylen Nightingale, PhD, MPH
Wake Forest School of Medicine
Medical Center Boulevard
Winston-Salem, NC 27157

However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.

By signing this form you give us permission to use your Protected Health Information for this study.

# WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or


Adult Consent Form



safety consequences. The investigators also have the right to stop your participation in the study at any time. This could be because we are unable to make contact with you or you have stopped providing care for your loved one.

You will be given any new information we become aware of that would affect your willingness to continue to participate in the study.

# WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or in the event of a research-related injury, contact the study investigator, Dr. Chandylen Nightingale.

The Institutional Review Board (IRB) is a group of people who review the research to protect your rights. If you have a question about your rights as a research participant, or you would like to discuss problems or concerns, have questions or want to offer input, or you want to obtain additional information, you should contact the Chairman of the IRB.

You will be given a copy of this signed consent form.

## **SIGNATURES**

I agree to take part in this study. I authorize the use and disclosure of my health information as described in this consent and authorization form. If I have not already received a copy of the Privacy Notice, I may request one or one will be made available to me. I have had a chance to ask questions about being in this study and have those questions answered. By signing this consent and authorization form, I am not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence.

| Subject Name (Printed): | | | |
|-------------------------------------|-------|-------|-------|
| Subject Signature: | Date: | Time: | am pm |
| Person Obtaining Consent (Printed): | | | |
| Person Obtaining Consent: | Date: | Time: | am pm |


Adult Consent Form